CLINICAL TRIAL: NCT03325959
Title: Hyperbaric Oxygen vs. Standard Pharmaceutical Therapies for Fibromyalgia Syndrome - Prospective, Randomized Crossover Clinical Trial
Brief Title: Hyperbaric Oxygen Compared to Pharmaceutical Therapies for Fibromyalgia Syndrome
Acronym: FMSRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0058-17-ASF
Record Dates: First submitted 2017-10-19; First posted 2017-10-30 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia; Hyperbaric Oxygen
Keywords: hyperbaric oxygen; HBOT; fibromyalgia; pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Hyperbaric Oxygenation; Therapeutics; Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial using conventional pharmacotherapy treatment compared to hyperbaric oxygen therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: randomization by computer, the patient and her primary care physician will know the treatment received. Any side effects during therapy will be reported to the care providers and nurses and physicians unrelated to the study. Investigators and outcome assessors will not know the patient's arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen therapy (Active Comparator): 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week. Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes Crossover: After 3 months of either pharmaceuitical or HBOT, once the 2nd evaluation is completed, all patients in both groups will be offered to switch to the alternative treatment group.
  Interventions: Device: Hyperbaric oxygen therapy (HBOT) treatment
- Pharmacotherapy (Active Comparator): patients will be offered pharmacological treatment with one of the two medications currently licensed for the treatment of FMS in Israel, i.e. Cymbalta and Lyrica. Treatment with Lyrica will start at a dose of 75 mg at bedtime while treatment with Cymbalta will start at a dose of 30 mg a day (in the morning). After a period of 6 weeks patients will be evaluated and dose will be adjusted as necessary. Patients may also be switched from one medication to the other based according to clinical judgment.
  Crossover: After 3 months of either pharmaceuitical or HBOT, once the 2nd evaluation is completed, all patients in both groups will be offered to switch to the alternative treatment group.
  Interventions: Drug: Cymbalta / Lyrica treatment; Device: Crossover Hyperbaric oxygen therapy

INTERVENTIONS:
Device: Hyperbaric oxygen therapy (HBOT) treatment — 60 HBOT sessions at 2 ATA 100% oxygen
  Arms: Hyperbaric oxygen therapy
Drug: Cymbalta / Lyrica treatment — one of the two medications currently licensed for the treatment of FMS in Israel, i.e. Cymbalta and Lyrica.
  Other Names: Cymbalta / Lyrica
  Arms: Pharmacotherapy
Device: Crossover Hyperbaric oxygen therapy — 60 HBOT sessions at 2 ATA 100% oxygen after crossover
  Arms: Pharmacotherapy

SUMMARY:
The investigators have previously studied the efficacy of hyperbaric oxygen therapy (HBOT) as a treatment for Fibromyalgia syndrome (FMS) in a prospective, active control, crossover clinical trial. The results demonstrated significant amelioration of all FMS symptoms, with significant improvement in life quality; furthermore, the investigators were able to demonstrate significant neuroplasticity on SPECT imaging, with a decrease of the hyperactivity in posterior regions and elevation of the reduced activity in frontal areas.

In the proposed study, the investigators intend to both repeat and expand our previous findings, treating FMS patients with HBOT while performing an extensive of evaluation both before and after treatment.

In the current study, the investigators plan to compare HBOT to current standard of care of FMS (pharmacological and non - pharmacological).

DETAILED DESCRIPTION:
The study will include 70 fibromyalgia patients in whom physical trauma, such mild traumatic brain injury (mTBI), could be considered as the trigger for FMS. Each participant will be examined at the time of recruitment and a diagnosis of FMS will be verified, based on the updated 2016 diagnostic criteria In the current study the investigators will recruit patients not currently being treated with medications specific for FMS, including anti-depression drugs, gabapentanoids and tricyclics, opiods and medical cannabis. Patients who are on such treatment will be required to discontinue treatment 2 weeks before recruitment.

Patients will undergo randomization upon recruitment to one of the two study groups. One group will proceed to a course of HBOT treatment while the second group will commence with standard treatment for FMS, as outlined in the Israeli guidelines for the diagnosis and treatment of FMS [41]. These patients will be given detailed education regarding the nature of FMS as well as recommendations regarding non - pharmacological interventions recommended for FMS, including graded physical exercise, hydrotherapy, movement-meditative treatments (e.g. Tai Chi) and cognitive behavioral treatment (CBT).

HBOT protocol: a total of 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week. 60 sessions will include exposure of 90 minutes to 100% at 2 Absolute atmospheres (ATA), with 5 minutes air breaks every 20 minutes.

Pharmaceutical protocol: patients will be offered pharmacological treatment with one of the two medications currently licensed for the treatment of FMS in Israel, i.e. Cymbalta and Lyrica. Treatment with Lyrica will start at a dose of 75 mg at bedtime while treatment with Cymbalta will start at a dose of 30 mg a day (in the morning). After a period of 6 weeks patients will be evaluated and dose will be adjusted as necessary. Patients may also be switched from one medication to the other based according to clinical judgment.

Crossover: After 3 months of either pharmaceuitical or HBOT, once the 2nd evaluation is completed, all patients in both groups will be offered to switch to the alternative treatment group.

ELIGIBILITY:
Inclusion Criteria:

* FMS diagnosis, based on the updated 2016 diagnostic criteria
* previous physical trauma (such as traumatic brain injury)

Exclusion Criteria:

* the presence of systemic inflammatory disorders including inflammatory rheumatological and autoimmune disorders.
* active malignancy,
* chronic ongoing infection
* major psychiatric disorders (excluding anxiety)
* Patients currently or previously treated with Duloxetine (Cymbalta) or Pregabalin (Lyrica) will also be excluded
* previous HBOT for any other reason prior to their inclusion;
* Chest pathology incompatible with pressure changes (including active asthma);
* Inner ear disease
* Claustrophobia;
* Inability to perform awake brain MRI test;
* Previous neurologic conditions (eg. Epilepsy, neuromuscular diseases, metabolic diseases, etc.);
* Brain tumors;
* Skull base fractures;
* s/p neurosurgery that included: ventricular drainage, subdural hematomas drainage, epidural hematomas drainage, intracerebral hemorrhage evacuation. Depressed fracture surgery, (Patients suffering from Encephalomalacia per MRI imaging will not be excluded).
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue Scale (VAS) | at 3 months
  The primary end point of the study will be the measurement of daily pain on a (0-10) Visual analogue Scale
Visual analogue Scale (VAS) | at 6 months
  The primary end point of the study will be the measurement of daily pain on a (0-10 scale) Visual analogue Scale

SECONDARY OUTCOMES:
Global Pain Scale (GPS) | baseline, at 3 months, at 6 months
  Fibromyalgia syndrome symptoms questionnaire named Global Pain Scale (GPS) questionnaire (0-100 scale)
Patient global impression of change | baseline, at 3 months, at 6 months
  Fibromyalgia syndrome symptoms questionnaire named: Patient global impression of change (yes/no)
Fibromyalgia Impact Questionnaire | baseline, at 3 months, at 6 months
  Fibromyalgia syndrome symptoms questionnaire named: Fibromyalgia Impact Questionnaire - FIQ (Hebrew version) (0-100 scale)
Wide Spread Pain Index | baseline, at 3 months, at 6 months
  Fibromyalgia syndrome symptoms questionnaire named:Wide Spread Pain Index (WPI) Fibromyalgia syndrome symptoms questionnaire named:Wide Spread Pain Index (scale 0-19)
Symptom Severity Scale | baseline, at 3 months, at 6 months
  Fibromyalgia syndrome symptoms questionnaire named:Symptom Severity Scale (SSS) (scale 0-12)
SF-36 questionnaire | baseline, at 3 months, at 6 months
  Quality of life questionnaire named short-form 36 (SF-36) (scale 0-100)
Medical Outcome Sleep Scale | baseline, at 3 months, at 6 months
  Sleep qualtiy questionnaire named: Medical Outcome Sleep Scale (MOS) questionnaire (0-100 scale)
Beck Depression Inventory | baseline, at 3 months, at 6 months
  Depression questionnaire named Beck Depression Inventory (BDI-II) (scale 0-63)
EQ-5D | baseline, at 3 months, at 6 months
  Quality of life questionnaire named EQ-5D (scale 0-25)
Cognitive function | baseline, at 3 months, at 6 months
  The Mindstreams battery includes several cognitive tests devised to check various aspects of brain capabilities. In the current study we will evaluate the cognitive indices based on the scores of the 6 cognitive tests listed below, which are expected to be relevant for mild TBI. For detailed description of all cognitive tests in Mindstreams battery
Cognitive function - CANTAB | baseline, at 3 months, at 6 months
  Patients' cognitive functions will be assessed by CANTAB computerized cognitive tests (Cambrdige cognition , England) [52]. The CANTAB is a semiautomated test battery which can be administered on a laptop PC and more recently has been modified for administration on a handheld tablet. The current release of CANTAB Eclipse comprises 25 tests designed to assess components of cognitive function which fall into 7 broad groups of tests: visual memory, executive function, working memory and planning, attention, semantic/verbal memory, decision making and response control, social cognition, and screening/familiarization.
Cerebral blood volume | baseline, at 3 months, at 6 months
  Cerebral blood volume (in mililiter) will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
  • DSC: 50 T2*-weighted gradient-echo echo planar imaging (EPI) volumes will be acquired, 2 repetitions before a bolus injection of Gadolinium-DTPA (Gd-DTPA), 48 repetitions after injection of Gd-DTPA.
Cerebral blood flow | baseline, at 3 months, at 6 months
  Cerebral blood volume (in mililiter/min) will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
  • DSC: 50 T2*-weighted gradient-echo echo planar imaging (EPI) volumes will be acquired, 2 repetitions before a bolus injection of Gadolinium-DTPA (Gd-DTPA), 48 repetitions after injection of Gd-DTPA.
Fractional anistropy | baseline, at 3 months, at 6 months
  Brain microstructure imaging will evalute fractional anistropy (FA , scale 0-1 in each region of interest. The MRI protocol will include diffusion tensor imaging (DTI).
  MRI sequence parameters:
  • DTI: 30 diffusion weighted images will be scanned with different gradient directions (b=1000) and one volume without diffusion weighting
Mean diffusivity | baseline, at 3 months, at 6 months
  Brain microstructure imaging will evalute mean diffusivity (MD, scale 0-1 in each region of interest. The MRI protocol will include diffusion tensor imaging (DTI).
  MRI sequence parameters:
  • DTI: 30 diffusion weighted images will be scanned with different gradient directions (b=1000) and one volume without diffusion weighting
Brain function imaging | baseline, at 3 months, at 6 months
  Resting state fMRI(rsfMRI or R-fMRI)- a method of functional brain imaging that can be used to evaluate regional interactions that occur when a subject is not performing an explicit task. This resting brain activity is observed through changes in blood flow in the brain which creates what is referred to as a blood-oxygen-level dependent (BOLD) signal that can be measured using functional Magnetic Resonance Imaging (fMRI).
brain function imaging | baseline, at 3 months, at 6 months
  Brain photon emission computed tomography (PET-CT) will be conducted using FDG.
Brain network analysis | baseline, at 3 months, at 6 months
  EEG activity will be recorded at resting state , during performing cognitive tasks and following a trans-magnetic stimulation. EEG recording will be performed using a 64 electrodes cap.
Heat/Cold Pain threshold evaluation | baseline, at 3 months, at 6 months
  Thermal pain is induced with thermal electrode (thermode). Thermode temperature will initially be set at 32.0°C and gradually increase at a rate of 0.3°C/sec. Participants will be instructed to report when the sensation produced by the thermode changed from heat sensation to pain (heat pain threshold) and when the pain became unbearable (heat pain tolerance). This procedure will be conducted twice for every subject and the mean of the two trials will be calculated. The thermode will be placed on adjacent areas of the forearm for every trial to avoid primary skin hyperalgesia.
Conditioned pain modulation | baseline, at 3 months, at 6 months
  In the current study CPM efficiency will be evaluated by computing the difference in mean pain intensity induced by the Heat test-stimulus (HTS) before and during immersion of non-dominant hand to 10 degrees cold water (the Cold pressor test) (i.e., pain during pre-immersion HTS - pain during post-immersion HTS). Thus, effective pain inhibitory mechanisms are represented by higher (positive) values.
Physical activity | baseline, at 3 months, at 6 months
  The daily physical activity will be objectively tracked by FitBit watch technology. The FitBit watch will be also wired during night for measurements of the time asleep, restless and awake, Fitbit trackers help you understand each night to make the most of each day
Exercise capacity | baseline, at 3 months, at 6 months
  Participants will undergo exercise testing using a modified Balke treadmill protocol and continuous expired gas analysis. Resting and exercise vital signs will monitored continuously. The exercise duration and exercise-limiting symptoms will be recorded. The peak VO2, VCO2 and respiratory exchange ratio (RER) will be averaged over the last 15 seconds of the exercise test. The ventilatory equivalent (VE/VCO2 slope) will be calculated from start of exercise to the end of exercise.
Inflammatory cytokines | baseline, at 3 months, at 6 months
  Blood Tests will include: IL-1, IL-6, Tumor necrosis factor-alpha, CRP.
CD4 number | baseline, at 3 months, at 6 months
  CD4 number (cells per ml) .Using a 4-color FACS CD4 number will be evaluated. Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
CD8 number | baseline, at 3 months, at 6 months
  CD8 number (cells per ml) .Using a 4-color FACS CD8 number will be evaluated. Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
CD4:CD8 ratio | baseline, at 3 months, at 6 months
  CD4:CD8 number (ratio) .Using a 4-color FACS CD4:CD8 number will be evaluated. Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
CD8+CD28null | baseline, at 3 months, at 6 months
  CD8+CD28null number (cells/ml) .Using a 4-color FACS CD8+CD28null number will be evaluated.
  Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
Naïve B-Cells number | baseline, at 3 months, at 6 months
  B cell number (cells/ml) .Using a 4-color FACS B cells number will be evaluated.
  Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
CD4CD25 positive number | baseline, at 3 months, at 6 months
  CD4CD25 cell number (cells/ml) .Using a 4-color FACS CD4CD25 number will be evaluated.
  Isolation of peripheral blood mononuclear cells (PBMC) will be isolated using density gradient centrifugation and will behed 3 times in 1640 RPMI medium. Cells will be frozen in freezing medium and kept in liquid nitrogen until thawed for analysis.
  PBMCs will be will behed twice in PBS with 3% FCS. 1X10^5 cells will be resuspended in 100 microliter PBS contatining CD4,CD8, CD25,CD28, CD56, CD16, CD3 conjugated colored antibodies.
Microbiome | baseline, at 3 months, at 6 months
  Microbiome evaluation method: Using our cutting-edge facilities, 16S ribosomal RNA (rRNA) next-generation sequencing of fecal samples will be performed to identify bacteria present in the gut. 16S rRNA gene sequencing is a well-established method for studying phylogeny and taxonomy (the description, identification and evolutionary classification) of samples from complex microbial environments that are difficult to study.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No